CLINICAL TRIAL: NCT04591561
Title: Incidence and Course of Stress Hyperglycemia in Critically Ill Children Admitted to PICU of Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Hamed Hussien, safaa.20124126@med.au.eau.eg, Assiut University
Other Study IDs: MRS in stress hyperglycemia
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stress Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detection of the prevelance of stress hyperglycemia in patients admitted to pediatric intensive care unit of Assiut university children hospital , asses its pattern ,course ,risk factors, its relation to the outcome and its management.

DETAILED DESCRIPTION:
Critically ill patients often develop endocrine and metabolic changes, particularly disruptions of glucose homeostasis that result in hyperglycemia and hypoglycemia.Stress hyperglycemia commonly occurs in children with critical illnesses.

Stress hyperglycemia results from increased gluconeogenesis relative to the clearance of glucose as well as from the development of insulin resistance affecting glucose uptake. These mechanisms are mediated through increased production of counteracting hormones (i.e., epinephrine, norepinephrine, cortisol, glucagon, and growth hormone). Furthermore, stress hyperglycemia is associated with pro-inflammatory cytokines, oxidative stress, and therapeutic interventions. Those factors in turn inhibit the secretion of insulin by pancreatic β cells through α-adrenergic receptor stimulation, interfere with insulin receptor signaling and/or insulin-regulated glucose channels, and directly interfere with proper glucose transport and utilization in peripheral cells.

Several studies have demonstrated the association of stress hyperglycemia in critically ill children with mortality. Specifically, peak and duration of stress hyperglycemia appear to be associated with mortality. Peak blood glucose concentrations tend to be much higher in non survivors compared with survivors. Similarly, non survivors tend to have exposure to longer duration of stress hyperglycemia compared with survivors. This association of stress hyperglycemia with mortality appears across different pediatric disease states, including septic shock, burns, traumatic brain injury, post cardiac surgery, and trauma. Additionally, stress hyperglycemia is associated with longer periods of ICU and hospital stay and more frequent nosocomial infections, including surgical site infections in critically ill children. While all these studies demonstrate strong associations between stress hyperglycemia and poor clinical outcomes, they do not necessarily demonstrate a cause and effect relationship.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill children admitted to emergency and intensive care unit with blood glucose level more than or equal 200 mg\dl.

Exclusion Criteria:

* Documented cases of diabetes mellitus

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with blood glucose above 200 mg/dl on admission to the emergency department will be considered to have hyperglycemia. Data will be collected . The blood sugar values will be followed up in these children until restoration of normoglycemia. All the children will be followed up till discharge or death in case of mortality
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of the prevelance of stress hyperglycemia in patients admitted to pediatric intensive care unit of Assiut university children hospital | baseline
  , asses its pattern ,course ,risk factors, its relation to the outcome and its management